CLINICAL TRIAL: NCT01438840
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial With an Open-label Extension Phase to Evaluate the Efficacy and Safety of Oral E5501 Plus Standard of Care for the Treatment of Thrombocytopenia in Adults With Chronic Immune Thrombocytopenia (Idiopathic Thrombocytopenia Purpura)
Brief Title: Efficacy and Safety of Oral E5501 Plus Standard of Care for the Treatment of Thrombocytopenia in Adults With Chronic Immune Thrombocytopenia (Amendment 02)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E5501-G000-302
Record Dates: First submitted 2011-09-19; First posted 2011-09-22 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Chronic Thrombocytopenia; Immune Thrombocytopenia
Keywords: Chronic Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Avatrombopag (Core Study) (Active Comparator): Avatrombopag will be administered orally as 5 mg, 10 mg, 20 mg, 30 mg, or 40 mg in a flexible dose design for 26 weeks. Participants will receive blinded therapy at a starting dose of 20 mg avatrombopag, one daily and allowed to have their dose titrated up (maximum dose of 40 mg avatrombopag) or down (minimum dose of 5 mg avatrombopag) depending on their response to study drug.
  Interventions: Drug: Avatrombopag; Drug: Standard of care
- Placebo (Core Study) (Placebo Comparator): Placebo will be administered as 5 mg, 10 mg, 20 mg, 30 mg or 40 mg in a flexible dose design for 26 weeks. Placebo will be administered orally at a starting dose of 20 mg, once daily. Afterwards the dose can be titrated up (maximum dose of 40 mg avatrombopag) or down (minimum dose of 5 mg avatrombopag) depending on the participant's response to the study drug; placebo titration will be used to maintain the blind.
  Interventions: Drug: Placebo; Drug: Standard of care
- Avatrombopag (Open-Label Extension) (Experimental): Participants who meet all eligibility criteria requirements of extension phase and who discontinue the core study because of lack of treatment effect will continue into the extension phase. Avatrombopag will be administered to participants who enter extension phase, with a starting dose of 20 mg avatrombopag, once daily for 76 weeks and undergo dose titration.
  Interventions: Drug: Avatrombopag; Drug: Standard of care

INTERVENTIONS:
Drug: Avatrombopag
  Other Names: E5501; Avatrombopag maleate
  Arms: Avatrombopag (Core Study); Avatrombopag (Open-Label Extension)
Drug: Placebo
  Arms: Placebo (Core Study)
Drug: Standard of care — Permitted ITP concomitant background therapies are as follows:
  * Corticosteroids and/or azathioprine taken at a stable dose for 4 weeks before randomization;
  * Mycophenolate mofetil (MMF) or danazol taken at a stable dose for at least 12 weeks before randomization;
  * Cyclosporine A (CsA) (due to the fact that it is a P-glycoprotein-mediated transport [P-gp] inhibitor) is to be avoided unless deemed medically necessary; CsA taken at a stable dose for at least 12 weeks before randomization.
  At the discretion of the investigator, participants will be allowed to use aspirin, other salicylates, or approved adenosine diphosphate (ADP) receptor antagonists, (eg, clopidogrel, prasugrel) during the study once their platelet count had risen.
  Participants treated with proton pump inhibitors (PPIs) and H2 antagonist therapy will receive a stable dose for at least 6 weeks prior to randomization. Treatment with these therapies must have been completed at least 2 weeks prior to randomization.

SUMMARY:
Core Study:

To demonstrate that the efficacy of avatrombopag (in addition to standard of care) is superior to placebo (in addition to standard of care) for the treatment of adult participants with chronic immune thrombocytopenia (idiopathic thrombocytopenic purpura) (ITP) as measured by cumulative number of weeks of platelet response over 6 months of once daily treatment in adults participants who received at least 1 prior ITP therapy.

Extension Phase:

To evaluate the safety and tolerability of long-term therapy with avatrombopag in participants with chronic ITP (cITP).

DETAILED DESCRIPTION:
This study consists three phases: Prerandomization, Randomization (Core Study) and Extension study. The overall duration of treatment (Core and Extension) is approximately 104 weeks with the Core study being 26 weeks and the Extension study being 76 weeks. Approximately 45 participants 18 years of age and over who meet all the eligibility requirements will be randomized. No single platelet count should be greater than 35x10^9/L (liter). Participants will be centrally stratified at randomization by splenectomy status, baseline platelet count, and use of concomitant ITP medication at baseline, and randomized to receive either double-blind avatrombopag or placebo in a 2:1 ratio. Participants will receive blinded therapy at a starting dose of 20 mg avatrombopag or placebo once daily. Participants will be allowed to have their dose titrated up (maximum dose 40 mg avatrombopag or matching placebo) or down (minimum dose 5 mg for avatrombopag or matching placebo) depending on their response to study drug. The goal of dose modification is to maintain the platelet count at levels greater than or equal to 50x10^9/L and less than or equal to 150x10^9/L, and to decrease the need for ITP-directed concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women greater than or equal to 18 years of age
2. Participants diagnosed with cITP (greater than or equal to 12 months duration) according to the American Society for Hematology/British Committee for Standards in Hematology (ASH/BCSH) guidelines, and an average of 2 platelet counts greater than 30x10^9/L). The physical exam should not suggest any disease which may cause thrombocytopenia other than ITP
3. Participants who previously received one or more ITP therapies (including, but not limited to corticosteroids, immunoglobulins, azathioprine, danazol, cyclophosphamide and/or rituximab).
4. Participants must have had either initially responded (platelet count greater than 50x10^9/L) to a previous ITP therapy or have had a bone marrow examination consistent with ITP within 3 years to rule out myelodysplastic syndrome (MDS) or other causes of thrombocytopenia
5. Prothrombin time/International Normalized Ratio (PT/INR) and activated partial thromboplastin time (aPTT) must have been within 80% to 120% of the normal range with no history of hypercoagulable state
6. A complete blood count within the reference range (including white blood count [WBC] differential not indicative of a disorder other than ITP), with the following exceptions: hemoglobin: participants with hemoglobin levels between 10 g/dL (100 g/L) and the lower limit of normal (LLN) are eligible for inclusion, if anemia was clearly attributable to ITP (excessive blood loss); Absolute neutrophil count (ANC) greater than or equal to 1500/uL (1.5x10^9/L) (elevated WBC/ANC due to corticosteroid treatment is acceptable)

Exclusion Criteria:

1. Participants with known secondary immune thrombocytopenia (e.g., with known Helicobacter pylori-induced ITP participants infected with known human immunodeficiency virus [HIV] or hepatitis C virus [HCV] or participants with known systemic lupus erythematosus). (Revised per Amendment 01)
2. Participants with significant medical conditions that may impact on the safety of the participant or interpretation of the study results (e.g., acute hepatitis, active chronic hepatitis; lymphoproliferative disease; myeloproliferative disorders, leukemia)
3. History of MDS
4. History of gastric atrophy (added per Amendment 01)
5. History of pernicious anemia or participants with vitamin B12 deficiency (defined as less than LLN) who have not had pernicious anemia excluded as a cause (added per Amendment 01)
6. Any prior history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), and more than two of the following risk factors: hormone replacement therapy, estrogen-containing hormone replacement or contraceptive therapies, smoking, diabetes, hypercholesterolemia, medication for hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, antithrombin III deficiency, etc.), or any other family history of arterial or venous thrombosis
7. Participants with a history of significant cardiovascular disease (e.g., congestive heart failure [CHF] New York Heart Association Grade III/IV, arrhythmia known to increase the risk of thromboembolic events [e.g., atrial fibrillation], participants with a QT interval corrected for heart rate of >450 msec, angina, coronary artery stent placement, angioplasty, coronary artery bypass grafting)
8. Participants with a history of cirrhosis, portal hypertension, and chronic active hepatitis
9. Participants with concurrent malignant disease
10. Use of immunoglobulins (IVIg and anti-D) within 1 week of randomization
11. Splenectomy or use of rituximab within 12 weeks of randomization
12. Use of romiplostim or eltrombopag within 4 weeks of randomization
13. Participants who are currently treated with corticosteroids or azathioprine but have not been receiving a stable dose for at least 4 weeks prior to randomization or have not completed these therapies more than 4 weeks prior to randomization
14. Participants who are currently treated with MMF, CsA, or danazol but have not been receiving a stable dose for at least 12 weeks prior to randomization or have not completed these therapies more than 4 weeks prior to randomization
15. Use of cyclophosphamide or vinca alkaloid regimens within 4 weeks of randomization
16. Participants who are currently treated with PPIs or H2 antagonist therapy but have not been receiving a stable dose for at least 6 weeks prior to randomization or have not completed these therapies more than 2 weeks prior to randomization
17. Fasting gastrin-17 blood levels exceeding the ULN at Screening for participants not on PPIs or H2 antagonists (Revised per Amendment 01)
18. Fasting gastrin-17 blood levels exceeding 1.5 times the upper limit of normal (ULN) at Screening for participants on PPIs or H2 antagonists (Added per Amendment 01)
19. Blood creatinine exceeding ULN by more than 20% OR total albumin below the lower limit of normal (LLN) by 10%
20. Alanine aminotransferase (ALT) OR aspartate aminotransferase (AST) levels exceeding 3 times the ULN or total bilirubin exceeding 2 times the ULN
21. Participants with a history of cancer treatment with cytotoxic chemotherapy and/or radiotherapy.
22. Participants with a history of ITP treatment with cytotoxic chemotherapy are still eligible for enrollment.
23. Females who are pregnant (positive beta-human chorionic gonadotropin positive [B-hCG] test) or breastfeeding
24. Participants with a known allergy to avatrombopag (E5501) or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02-16 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe McIntosh, Study Director — Eisai Inc.
Locations (25):
- Australia (2):
  - Adelaide
  - Bedford Park
- Antwerp, Belgium
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- Rotterdam, Netherlands
- New Zealand (2):
  - Christchurch
  - Palmerston North
- Poland (6):
  - Bialystok
  - Chorzów
  - Gdansk
  - Krakow
  - Lodz
  - Wroclaw
- Singapore, Singapore
- Bratislava, Slovakia
- Johannesburg, South Africa
- Ukraine (5):
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kyiv
  - Lviv

REFERENCES:
- [Derived] Jurczak W, Chojnowski K, Mayer J, Krawczyk K, Jamieson BD, Tian W, Allen LF. Phase 3 randomised study of avatrombopag, a novel thrombopoietin receptor agonist for the treatment of chronic immune thrombocytopenia. Br J Haematol. 2018 Nov;183(3):479-490. doi: 10.1111/bjh.15573. Epub 2018 Sep 7. PMID 30191972

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 100 participants were screened in study. Of these 100 participants, 51 were screen failures and 49 were randomized into the study.
Groups:
- Placebo (Core Study): Placebo was administered as 5 mg, 10 mg, 20 mg, 30 mg or 40 mg in a flexible dose design for 26 weeks. Placebo was administered orally at a starting dose of 20 mg, once daily. Afterwards the dose could be titrated up (maximum dose of 40 mg avatrombopag) or down (minimum dose of 5 mg avatrombopag) depending on the participant's response to the study drug; placebo titration was used to maintain the blind.
- Avatrombopag (Core Study): Avatrombopag was administered orally as 5 mg, 10 mg, 20 mg, 30 mg, or 40 mg in a flexible dose design for 26 weeks. Participants received blinded therapy at a starting dose of 20 mg avatrombopag, one daily and they were allowed to have their dose titrated up (maximum dose of 40 mg avatrombopag) or down (minimum dose of 5 mg avatrombopag) depending on their response to study drug.
- Avatrombopag (Extension Phase): Participants who met all the eligibility criteria requirements of extension phase and who discontinued the core study because of lack of treatment effect continued into the extension phase. Avatrombopag was administered to participants who entered extension phase, with a starting dose of 20 mg avatrombopag, once daily for 76 weeks and underwent dose titration.
Period: Core Study
Arm/Group | Placebo (Core Study) | Avatrombopag (Core Study) | Avatrombopag (Extension Phase)
Started | 17 | 32 | 0
Completed | 1 | 22 | 0
Not Completed | 16 | 10 | 0
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Lack of Efficacy | 15 | 7 | 0
Not completed — Withdrawal of consent | 1 | 0 | 0
Period: Extension Phase
Arm/Group | Placebo (Core Study) | Avatrombopag (Core Study) | Avatrombopag (Extension Phase)
Started | 0 | 0 | 39 (39 participants met eligibility criteria for the Extension Phase.)
Completed | 0 | 0 | 29
Not Completed | 0 | 0 | 10
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Core Study) | Avatrombopag (Core Study) | Total
Number analyzed (Participants) | 17 | 32 | 49
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 41.2 (14.7) | 46.4 (14.2) | 44.6 (14.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 23 | 31
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Weeks With Platelet Count Greater Than or Equal to 50 x 10^9/L During 6-Month Treatment Period
Description: The cumulative number of weeks of platelet response is defined as the total numbers of weeks in which the platelet count is greater than or equal to 50 x 10^ 9/L during 6 months of treatment of core study in the absence of rescue therapy.
Time Frame: Week 1 to Week 26
Population: Full Analysis Set (Core Study): All participants who were randomized into the study.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Placebo (Core Study) | Avatrombopag (Core Study)
Number analyzed (Participants) | 17 | 32
Weeks | 0 [0 to 2] | 12.4 [0 to 25]
Statistical Analysis 1: Comparison: Placebo (Core Study) vs Avatrombopag (Core Study); Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants With a Reduction in Use of Concomitant Immune/Idiopathic Thrombocytopenic Purpura (ITP) Medication
Description: Only participants on concomitant ITP medications at baseline were included.
Time Frame: Week 1 through Week 26
Population: Full Analysis Set (Core Study): All participants who were randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Core Study) | Avatrombopag (Core Study)
Number analyzed (Participants) | 7 | 15
Participants
  Yes | 0 | 5
  No | 7 | 10

3. Secondary Outcome: Number of Participants With Platelet Count Greater Than or Equal to 50 x 10^9/L at Day 8
Description: Participants with platelet response at Day 8 are defined as those who had a platelet count greater than or equal to 50 x 10^9/L at day 8 in the absence of rescue therapy on or before Day 8.
Time Frame: Week 1 (Day 8)
Population: Full Analysis Set (Core Study): All participants who were randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Core Study) | Avatrombopag (Core Study)
Number analyzed (Participants) | 17 | 32
Participants
  Yes | 0 | 21
  No | 17 | 11

ADVERSE EVENTS:
Time Frame: Core Study: up to 39 Weeks (including Screening, Titration, Treatment, Dose Taper, and Follow-up for those who did not enter the Extension Phase). Extension Phase: up to 104 weeks (including Conversion, Maintenance Period, Dose Taper, and Follow-up).
Description: Treatment emergent adverse events were collected. Core Study Safety Analysis Set (SAS): All participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment. Extension Phase SAS: All participants who received at least 1 dose of avatrombopag (either Core or Extension Phase) and had a postdose safety assessment.
Groups:
- Avatrombopag (Extension Phase): Participants who met all eligibility criteria requirements of extension phase and who discontinued the core study because of lack of treatment effect continued into the extension phase. Avatrombopag was administered to participants who entered extension phase, with a starting dose of 20 mg avatrombopag, once daily for 76 weeks and underwent dose titration.
Arm/Group | Placebo (Core Study) | Avatrombopag (Core Study) | Avatrombopag (Extension Phase)
Serious Adverse Events (participants affected / at risk) | 1/17 | 9/32 | 15/47
Other Adverse Events (participants affected / at risk) | 10/17 | 31/32 | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Core Study) (N=17) | Avatrombopag (Core Study) (N=32) | Avatrombopag (Extension Phase) (N=47)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Polyserositis (General disorders) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Core Study) (N=17) | Avatrombopag (Core Study) (N=32) | Avatrombopag (Extension Phase) (N=47)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 4 | 8
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 3 | 4
Nausea (Gastrointestinal disorders) | 0 | 3 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Fatigue (General disorders) | 1 | 4 | 7
Influenza (Infections and infestations) | 0 | 2 | 4
Nasopharyngitis (Infections and infestations) | 0 | 3 | 5
Pharyngitis (Infections and infestations) | 1 | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 6 | 11
Urinary tract infection (Infections and infestations) | 0 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 4 | 10 | 19
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood gastrin increased (Investigations) | 0 | 2 | 2
Blood urine present (Investigations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 2 | 12 | 14
Somnolence (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 8
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 4 | 7
Hypertension (Vascular disorders) | 1 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other